CLINICAL TRIAL: NCT07313254
Title: Clinical And Radiographic Evaluation Of Zinc Substituted Nanohyrdoxyappatite Bone Graft And Advanced Platelet Rich Fibrin Block In The Treatment Of Periodontal Intrabony Defects: A Randomized Controlled Study
Brief Title: Clinical And Radiographic Evaluation Of Zinc Substituted Nanohyrdoxyappatite Bone Graft And Advanced Platelet Rich Fibrin Block In The Treatment Of Periodontal Intrabony Defects
Acronym: R C S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 596/2022
Record Dates: First submitted 2025-08-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis; Periodontal Diseases
Keywords: nano-hydroxyapatite; advanced platelet-rich fibrin blocks; zinc-substituted nano-hydroxyapatite
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- treating with zinc substituted hydroxyapatite graft combined with PRF block using full flap (Active Comparator): patients were treated with zinc substituted hydroxyapatite graft combined with platelet rich fibrin block using a full thickness mucoperiosteal flap surgical technique.
  After the pretreatment phase, patients were recalled under local anesthesia an intrasulcular incision was performed with #15 blade elevating a full-thickness mucoperiosteal flap and after removing all the inflammatory granulation tissue we put in the defect Zinc substituted nano-hydroxyapatite graft combined in platelet-rich fibrin block (A-PRF +I-PRF+graft ).
  Zinc substituted nano hydroxyapatite graft was taken in a bone well, to which i-PRF was mixed and the cut pieces of the A-PRF membrane were incorporated. The resulted cohesive, packable graft "PRF block" which were placed into the defect.
  Then the mucoperiosteal flap returned to its position in both groups and sutured using silk suture size (4/0).
  Interventions: Procedure: OFD with zinc substituted nano HA combined with PRF block
- treating with zinc substituted nano-hydroxyapatite graft using a full thickness mucoperiosteal flap (Active Comparator): patients were treated with zinc substituted nano-hydroxyapatite graft using a full thickness mucoperiosteal flap surgical technique.
  Interventions: Procedure: OFD with zinc substituted nano HA
- treating with a nano-hydroxyapatite graft using full thickness mucoperiosteal flap surgical techniq (Active Comparator): patients were treated with a nano-hydroxyapatite graft using a full thickness mucoperiosteal flap surgical technique.
  Interventions: Procedure: OFD with nano HA

INTERVENTIONS:
Procedure: OFD with zinc substituted nano HA combined with PRF block — After the pretreatment phase, patients were recalled under local anesthesia an intrasulcular incision will performed with #15 blade elevating a full-thickness mucoperiosteal flap and after removing all the inflammatory granulation tissue we put in the defect Zinc substituted nano-hydroxyapatite graft combined in platelet-rich fibrin block (A-PRF +I-PRF+graft ). Zinc substituted nano hydroxyapatite graft was taken in a bone well, to which i-PRF was mixed and the cut pieces of the A-PRF membrane were incorporated. The resulted cohesive, packable graft "PRF block" which were placed into the defect. Then the mucoperiosteal flap returned to its position in both groups and sutured using silk suture size (4/0).
  Arms: treating with zinc substituted hydroxyapatite graft combined with PRF block using full flap
Procedure: OFD with zinc substituted nano HA — After the pretreatment phase, patients were recalled under local anesthesia an intrasulcular incision will performed with #15 blade elevating a full-thickness mucoperiosteal flap and after removing all the inflammatory granulation tissue we put in the defect Zinc substituted nano-hydroxyapatite graft. Then the mucoperiosteal flap returned to its position in both groups and sutured using silk suture size (4/0).
  Arms: treating with zinc substituted nano-hydroxyapatite graft using a full thickness mucoperiosteal flap
Procedure: OFD with nano HA — After the pretreatment phase, patients were recalled under local anesthesia an intrasulcular incision will performed with #15 blade elevating a full-thickness mucoperiosteal flap and after removing all the inflammatory granulation tissue we put in the defect nano-hydroxyapatite graft Then the mucoperiosteal flap returned to its position in both groups and sutured using silk suture size (4/0).
  Arms: treating with a nano-hydroxyapatite graft using full thickness mucoperiosteal flap surgical techniq

SUMMARY:
Periodontal intrabony defects pose a significant challenge in clinical dentistry due to their complex anatomy and limited regenerative potential. Recent advancements in biomaterials and regenerative techniques have introduced novel approaches to enhance periodontal healing. This study evaluates the clinical and radiographic outcomes of using nano-hydroxyapatite (nHA) and zinc-substituted nano-hydroxyapatite (Zn-nHA) in combination with advanced platelet-rich fibrin (A-PRF) blocks for the treatment of periodontal intrabony defects.

Nano-hydroxyapatite, a biomimetic material, has shown promise in promoting bone regeneration due to its osteoconductive properties. Zinc substitution further enhances its biological activity by incorporating antimicrobial and osteoinductive characteristics. Advanced PRF, a second-generation platelet concentrate, provides a scaffold rich in growth factors and cytokines, which synergistically supports tissue regeneration.

DETAILED DESCRIPTION:
Periodontitis causes deep periodontal pockets due to bone and attachment loss. Zinc-substituted hydroxyapatite enhances bone regeneration, while PRF promotes healing through growth factors. Their combination as a PRF block offers a promising approach for periodontal defect repair. This randomized controlled clinical trial was conducted to compare the effectiveness of zinc-substituted nano-hydroxyapatite alone and in combination with platelet-rich fibrin (PRF) block in the treatment of intrabony periodontal defects. Thirty patients diagnosed with periodontitis were selected based on defined inclusion and exclusion criteria and were randomly allocated into three equal groups. Each group received a different grafting material using a full-thickness mucoperiosteal flap surgical technique. Standardized clinical parameters-including gingival index, plaque index, probing pocket depth, and clinical attachment level-were recorded at baseline and six months post-operatively. Radiographic assessments were also performed to evaluate bone changes using digital imaging and image analysis software. The zinc-substituted grafts were prepared using a chemical process, and PRF blocks were created by combining advanced and injectable PRF with the graft material

ELIGIBILITY:
Inclusion Criteria:

1. Adequate oral hygiene conditions.
2. Age range from 20 years to 50 years.
3. All patients will be physically healthy.
4. Patients who are co-operatively motivated.

Exclusion Criteria:

1. Those who smoke.
2. Women who are pregnant.
3. Patients with poorly controlled systemic diseases which preclude local anesthesia or surgical procedures.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
measurement of gingival indices | From enrollment to the end of treatment at 6 months
  Gingival index (Loe et al.,1963):
  Score Criteria:
  0- No inflammation.
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
measurement of plaque indices | 6 monthes
  • Plaque index (Silness et al.,1964):
  We determine the amount of plaque on the tooth surface using a scale from 0 to 3:
  0- No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth, which could not be seen with the naked eye. But only by using disclosing solutions or by using probe.
  2. Moderate accumulation of deposits within the gingival pocket, on the gingival margin and/ or adjacent tooth surface, which could be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
measurement of probing pocket depth | 6 months
  Probing pocket depth :
  Probing pocket depth (PD) is measured by using William's graduated probe from the free gingival margin to the base of the periodontal pocket.
Measurement of Clinical attachment level | 6 months
  The clinical attachment level (CAL) is measured by using periodontal probe from the cemento - enamel junction to the bottom of the pocket at each selected site.

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Yehia, Ismailia, Ismailia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet

REFERENCES:
- [Result] Bhardwaj VA, Deepika PC, Basavarajaiah S. Zinc Incorporated Nano Hydroxyapatite: A Novel Bone Graft Used for Regeneration of Intrabony Defects. Contemp Clin Dent. 2018 Jul-Sep;9(3):427-433. doi: 10.4103/ccd.ccd_192_18. PMID 30166839
- See also: Zinc Incorporated Nano Hydroxyapatite: A Novel Bone Graft Used for Regeneration of Intrabony Defects — https://pmc.ncbi.nlm.nih.gov/articles/PMC6104351/